CLINICAL TRIAL: NCT06560476
Title: A Prospective Multi-site Registry of Real-world Experience With the OPtilume™ BPH Catheter SystEm for Treatment of Men eXperiencing Symptomatic BPH
Brief Title: OPtilume™ BPH Catheter SystEm for Treatment of Men eXperiencing Symptomatic BPH
Acronym: APEX
Status: Recruiting | Type: Observational
Sponsor: Urotronic Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR1326
Record Dates: First submitted 2024-06-20; First posted 2024-08-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH; Drug Coated Balloon; DCB; Prostate; LUTS; Optilume
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Arm: This is the data collection study arm. There is no other arm in the study.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Subject's data will be collected from patients that are undergoing care using the Optilume drug-coated catheter system.

SUMMARY:
APEX is a prospective multi-site registry of real-world experience with the Optilume™ BPH Catheter System for treatment of men experiencing symptomatic BPH.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated with the Optilume BPH Catheter System in accordance with the Instructions for Use (IFU).

Exclusion Criteria:

1. Unwilling to abstain from sexual intercourse or use a condom for 30 days post-procedure and utilize a highly effective contraceptive for at least 12 months post-procedure
2. Presence of an artificial urinary sphincter, penile prosthesis, or stent(s) in the urethra or prostate
3. Confirmed or suspected malignancy of prostate or bladder.
4. Active urinary tract infection (UTI)
5. Anatomy (e.g., presence of false passage or size of meatus) is not suitable for treatment with the Optilume BPH Catheter System

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Must be a male
Study Population: Men experiencing symptomatic BPH that are seeking the Optilume drug coated catheter system.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the average IPSS change from baseline to 12 months. | Baseline to 12 months
  The primary efficacy endpoint is the average IPSS change from baseline to 12 months.
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms.
  It is a validated, reproducible scoring system to assess disease severity and response to therapy.
  The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
  It is not a reliable diagnostic tool for lower urinary tract symptoms (LUTS) suggestive of BPH, but can be used to quantitatively measure LUTS after a diagnosis is made.
The primary safety endpoint is the freedom from treatment-related adverse SAEs. | Baseline to 12 months
  The primary safety endpoint is the freedom from treatment-related adverse SAEs.

SECONDARY OUTCOMES:
Frequency and severity of treatment-related AEs | From baseline to through study completion, an average of 2 years.
  Adverse events will be collected and assessed for relatedness to the device and the procedure as well as for severity. The Clavien-Dindo severity grading scale is a commonly used criteria in the urology community.
Change in IPSS over time | From baseline to through study completion, an average of 2 years.
  The IPSS tool is the most commonly reported symptom score for obstructive urinary symptoms secondary to BPH. Average IPSS scores, absolute change from baseline, and percent change from baseline will be reported at each follow-up timepoint.
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms.
  It is a validated, reproducible scoring system to assess disease severity and response to therapy.
  The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
  It is not a reliable diagnostic tool for lower urinary tract symptoms (LUTS) suggestive of BPH, but can be used to quantitatively measure LUTS after a diagnosis is made.
Change in Qmax (mL per second) over time | From baseline to through study completion, an average of 2 years.
  Uroflowmetry represents an objective measure of relief of obstruction. Average peak urinary flow rate (Qmax) and change from baseline will be reported at each follow-up timepoint.
  Uroflowmetry assesses flow pattern, flow curve shape, maximum urinary flow (Qmax), voided volume (VV), voiding time (VT), PVR volume (PVR). A minimum of 150ml is required to provide an accurate assessment in men
Change in PVR over time | From baseline to through study completion, an average of 2 years.
  Residual urine in the bladder due to incomplete emptying is an important clinical consideration in subjects with obstructive BPH. Average PVR and change from baseline will be reported at each follow-up timepoint.
  Post-void residual volume (PVR) is the amount of urine retained in the bladder after a voluntary void and functions as a diagnostic tool. A PVR can be used to assess many disease processes, including but not limited to neurogenic bladder, cauda equina syndrome, urinary outlet obstruction, mechanical obstruction, medication-induced urinary retention, postoperative urinary retention, and urinary tract infections. The PVR may be determined through urinary catheterization, a portable dedicated bladder scanner, or a formal ultrasound examination.
Freedom from repeat intervention (time-to-event) | From baseline to through study completion, an average of 2 years.
  The proportion of subjects free from repeat surgical or endoscopic intervention for BPH will be reported over time utilizing the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Golden State Urology, Sacramento, California
  - Florida Urology Partners, Tampa, Florida
  - Kearney Urology Center, Kearney, Nebraska
  - The Urology Center, P.C., Omaha, Nebraska
  - Sheldon Freedman, Ltd, Las Vegas, Nevada
  - Northwell Health - Smith Institute of Urology, Syosset, New York
  - Good Samaritan Hospital, Corvallis, Oregon
  - Midtown Urology, Austin, Texas
  - Potomac Urology, Woodridge, Virginia

IPD SHARING:
Plan to Share IPD: No